CLINICAL TRIAL: NCT06994325
Title: A Pilot Hybrid Effectiveness-Implementation Trial for the Conversations Helpful for Awareness of Illness Trajectory (CHAT) Intervention
Brief Title: Testing the CHAT Program for Patients With Heart Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-07027766; 1R21AG077092-01A1 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: HFpEF; CHAT; Conversations Helpful for Awareness of Illness Trajectory; Effectiveness-Implementation Trial; Heart Failure with Preserved Ejection Fraction
MeSH Terms: interventions — Methods; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Group (Active Comparator): Subjects randomized to the standard of care group will receive usual care (and will not receive the CHAT intervention).
  Interventions: Behavioral: Standard of Care (SOC)
- CHAT Intervention Group (Experimental): The group randomized to the CHAT intervention will be instructed to watch 7 short patient-facing videos and participate in four biweekly sessions with a trained health coach.
  Interventions: Behavioral: Conversations Helpful for Awareness of Illness Trajectory (CHAT) Intervention

INTERVENTIONS:
Behavioral: Conversations Helpful for Awareness of Illness Trajectory (CHAT) Intervention — The Conversations Helpful for Awareness of illness Trajectory (CHAT) intervention will incorporate 4 health-coach sessions, supplemented by 7 educational videos. Each session will be up to 60 minutes long and will be conducted remotely. During the health coach sessions, a trained health coach will work with subjects, reviewing the content of each video and emphasizing key learning content.
  Arms: CHAT Intervention Group
Behavioral: Standard of Care (SOC) — The Standard of Care Group will not have access to the Health Coach or video-based educational content. This group will have no study activities during Weeks 1-7 but will participate in follow-up assessments.
  Arms: Standard of Care Group

SUMMARY:
The researchers are studying whether an intervention that involves video-based educational content and a health coach is acceptable, feasible, and effective for people with Heart Failure with Preserved Ejection Fraction (HFpEF).

DETAILED DESCRIPTION:
This is a pilot randomized controlled trial of 50 subjects that will compare the CHAT intervention (video-based educational content and a health coach) with usual care. Video-based educational content was developed based on Adult Learning Theory and Social Cognitive Theory. Key content areas covered by the videos and health coach will include: HFpEF Overview, Signs and Symptoms of HFpEF, Medication Management, Physical Activity and Diet with HFpEF, and Planning for the Future (Advance Care Planning).

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female ≥ 60 years old
2. Documentation of HFpEF according to clinical practice guidelines (signs & symptoms of HF AND ejection fraction ≥50%)

Exclusion Criteria:

1. Previously referred to hospice care
2. Prior completion of advance directives
3. Moderate-severe dementia or psychiatric disorder precluding informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline on the Self-Care of Heart Failure Index (SCHFI) Summary Score at 90 Days | Baseline, 90 days
  This measure uses the SCHFI, a 29-item survey that evaluates three subscales: Symptom Perception, Self-Care Management, and Self-Care Maintenance, with the lowest possible score of 0 and the highest possible score of 100. Higher scores indicate better self-care. Standardized scoring will assess changes from baseline.

SECONDARY OUTCOMES:
Scores on the Feasibility of Intervention Measure (FIM) at 90 Days | 90 days
  This metric uses the FIM, a 4-item survey rated on a 5-point Likert scale, where the lowest score of 1 indicates 'completely disagree' and the highest score of 5 indicates 'completely agree'. Higher scores suggest greater perceived feasibility of the CHAT intervention.
Scores on the Intervention Appropriateness Measure (IAM) at 90 Days | 90 days
  This measure uses the IAM, a 4-item survey rated on a 5-point Likert scale, where the lowest score of 1 indicates 'completely disagree' and the highest score of 5 indicates 'completely agree'. The IAM assesses perceived appropriateness of the CHAT intervention. Higher scores suggest better perceived alignment with patient needs.
Scores on the Acceptability of Intervention Measure (AIM) at 90 Days | 90 days
  This measure uses the AIM, a 4-item survey rated on a 5-point Likert scale, where the lowest score of 1 indicates 'completely disagree' and the highest score of 5 indicates 'completely agree'. The AIM evaluates participants' perceptions of the CHAT intervention's acceptability. Higher scores suggest better acceptance by participants.
Mean Change from Baseline on the Advance Care Planning Engagement Survey at 90 Days | Baseline, 90 days
  This metric assesses engagement in Advance Care Planning (ACP) using a 4-item survey rated on a 5-point Likert scale, where the lowest score of 1 indicates 'I have never thought about it ' and the highest score of 5 indicates 'I have already done it'. The mean score is calculated, with higher scores indicating increased engagement in ACP.
Mean Change from Baseline on the Advance Care Planning Readiness Scale at 90 Days | Baseline, 90 days
  This metric assesses readiness in Advance Care Planning (ACP) using an 8-item survey rated on a 7-point Likert scale, where the lowest score of 1 indicates 'strongly disagree' and the highest score of 7 indicates 'strongly agree'. The mean score is calculated, with higher scores indicating increased readiness in ACP.
Mean Change from Baseline for Percentage of Participants Completing a Health Care Proxy Form at 90 days | Baseline, 90 days
  This measure uses the Advance Directive Completion Question to count the number of participants who complete a health care proxy form, out of the number of total study participants, reflecting their engagement in Advance Care Planning.
Mean Change from Baseline for Percentage of Participants Completing a Living Will Form at 90 days | Baseline, 90 days
  This measure uses the Advance Directive Completion Question to count the number of participants who complete a living will form, out of the number of total study participants, reflecting their involvement in planning for future healthcare decisions.
Mean Change from Baseline on the Perceived Health Competency Scale (PHCS) at 90 Days | Baseline, 90 days
  The PHCS is an 8-item survey, rated on a 5-point Likert scale, where the lowest score of 1 indicates 'strongly disagree' and the highest score of 5 indicates 'strongly agree'. Scores are calculated by summing item responses, with higher scores indicating greater perceived ability to manage health.
Mean Change from Baseline on the Patient Activation Measure (PAM) at 90 Days | Baseline, 90 days
  The PAM is a 10-item survey, rated on a 4-point Likert scale, where the lowest score of 1 indicates 'disagree strongly' and the highest score of 4 indicates 'agree strongly'. Scores are calculated by summing item responses and converting them to an overall activation level, with higher scores indicating greater self-management and engagement in health.
Mean Change from Baseline on The Human Connection (THC) Scale at 90 Days | Baseline, 90 days
  The Human Connection (THC) Scale measures therapeutic alliance with 16 items rated on a 4-point Likert scale, with the lowest possible score of 1 and the highest possible score of 4. The mean score reflects perceived improvements in the therapeutic relationship.
Mean Change from Baseline on the Basic Psychological Need Satisfaction and Frustration Scale (BPNSF) Relatedness Subscale at 90 Days | Baseline, 90 days
  This measure uses the Relatedness Subscale of the BPNSF, an 8-item survey rated on a 5-point Likert scale, where the lowest score of 1 indicates 'completely disagree' and the highest score of 5 indicates 'completely agree'. The BPNSF assesses perceived satisfaction and frustration in relationships. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Parag Goyal, MD, MSc, Principal Investigator — Weill Medical College of Cornell University; Megan J Shen, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the CHAT study will be shared only after the publication of findings addressing the study's specific aims. Data generated under this project will be managed in accordance with the policies of Weill Cornell Medicine (WCM) and the NIH, including the NIH Data Sharing Policy and Implementation Guidance. After publication of our main findings, data will be made available for secondary analyses. External researchers may request access to the data by submitting a written proposal outlining the hypotheses to be tested. All data will be de-identified to protect participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be shared after we have published the specific aims of this study. There is no end date to access the data from the research project.
Access Criteria: Researchers granted access to the data will be required to use it solely for research purposes, ensuring that no individual participants are identifiable. They must also implement appropriate security measures, such as using password-protected servers and files, to safeguard the data. Upon completion of the analyses, the data must be returned or destroyed. Released datasets will be subject to stringent safeguards to ensure compliance with the Health Insurance Portability and Accountability Act (HIPAA). Additionally, a data-sharing agreement will be required, specifying that the data is used exclusively for research purposes and that no participants are identifiable. A data management plan will also be necessary to ensure the continued security and confidentiality of the data, as well as to outline the process for returning or destroying the data once the analysis is complete.

REFERENCES:
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW; ACC/AHA Joint Committee Members. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 May 3;145(18):e895-e1032. doi: 10.1161/CIR.0000000000001063. Epub 2022 Apr 1. PMID 35363499
- [Background] Jankowska A, Mlynczak K, Golicki D. Validity of EQ-5D-5L health-related quality of life questionnaire in self-reported diabetes: evidence from a general population survey. Health Qual Life Outcomes. 2021 May 5;19(1):138. doi: 10.1186/s12955-021-01780-2. PMID 33952271
- [Background] Spertus JA, Jones PG. Development and Validation of a Short Version of the Kansas City Cardiomyopathy Questionnaire. Circ Cardiovasc Qual Outcomes. 2015 Sep;8(5):469-76. doi: 10.1161/CIRCOUTCOMES.115.001958. PMID 26307129
- [Background] Chen B, Vansteenkiste M, Beyers W, et al. Basic Psychological Need Satisfaction and Frustration Scale. Motivation and Emotion. 2015;
- [Background] Mack JW, Block SD, Nilsson M, Wright A, Trice E, Friedlander R, Paulk E, Prigerson HG. Measuring therapeutic alliance between oncologists and patients with advanced cancer: the Human Connection Scale. Cancer. 2009 Jul 15;115(14):3302-11. doi: 10.1002/cncr.24360. PMID 19484795
- [Background] Riegel B, Lee CS, Dickson VV, Carlson B. An update on the self-care of heart failure index. J Cardiovasc Nurs. 2009 Nov-Dec;24(6):485-97. doi: 10.1097/JCN.0b013e3181b4baa0. PMID 19786884
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Brown AJ, Shen MJ, Urbauer D, Taylor J, Parker PA, Carmack C, Prescott L, Rosemore C, Kolawole E, Sun C, Ramondetta L, Bodurka DC. The Advance Care Planning Readiness Scale: Development and Validation of a Measure of Willingness to Discuss and Acceptance of End-of-Life Care in Gynecologic Cancer Patients. Int J Gynecol Cancer. 2017 May;27(4):838-846. doi: 10.1097/IGC.0000000000000953. PMID 28399031
- [Background] Sudore RL, Stewart AL, Knight SJ, McMahan RD, Feuz M, Miao Y, Barnes DE. Development and validation of a questionnaire to detect behavior change in multiple advance care planning behaviors. PLoS One. 2013 Sep 5;8(9):e72465. doi: 10.1371/journal.pone.0072465. eCollection 2013. PMID 24039772
- [Background] Riegel B, Barbaranelli C, Carlson B, Sethares KA, Daus M, Moser DK, Miller J, Osokpo OH, Lee S, Brown S, Vellone E. Psychometric Testing of the Revised Self-Care of Heart Failure Index. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):183-192. doi: 10.1097/JCN.0000000000000543. PMID 30303894